CLINICAL TRIAL: NCT05334004
Title: A Phase I Study of Intra-anally Administered Lopinavir/Ritonavir in People Living With HIV (PLWH) With High-Grade Anal Intraepithelial Neoplasia (AIN 2/3)
Brief Title: Lopinavir/Ritonavir in PLWH With High-Grade AIN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Wisconsin Partnership Program (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2023-0052; SMPH/SURGERY/COLON RECT (Other: UW Madison); Protocol Version 12/23/25 (Other: UW Madison); 2022-0468 [former] (Other: UW Madison); UW22123 (Other: UWCCC ID)
Record Dates: First submitted 2022-04-01; First posted 2022-04-19 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-05

CONDITIONS: High-Grade Anal Intraepithelial Neoplasia
MeSH Terms: interventions — Lopinavir

STUDY DESIGN:
Intervention Model Description: modified 3+3 design with increasing concentrations of study drug and thorough assessment of potential toxicities.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Cohort 1: Lopinavir/Ritonavir 200mg/50mg (2 cycles) (Experimental): Cohort 1 will receive two 5-day cycles of the low dose of the suppository (Lopinavir/Ritonavir (200mg/50mg)) in Weeks 0 and 2
  Interventions: Drug: Lopinavir / Ritonavir
- Cohort 1b: Lopinavir/Ritonavir 200mg/50mg (3 cycles) (Experimental): Cohort 1b will receive three 5-day cycles of the low dose of the suppository (Lopinavir/Ritonavir (200mg/50mg)) in Weeks 0, 2, and 4 if Cohort 2 has one dose-limiting toxicity (DLT).
  Interventions: Drug: Lopinavir / Ritonavir
- Cohort 2: Lopinavir/Ritonavir 400mg/100mg (2 cycles) (Experimental): Cohort 2 will receive two 5-day cycles of the higher dose of the suppository (Lopinavir/Ritonavir (400mg/100mg)) in Weeks 0 and 2, if Cohort 1 dose is safe.
  Interventions: Drug: Lopinavir / Ritonavir
- Cohort 2b: Lopinavir/Ritonavir 400mg/100mg (3 cycles) (Experimental): Cohort 2b will receive three 5-day cycle of the higher dose of the suppository (Lopinavir/Ritonavir (400mg/100mg)) in Weeks 0, 2 and 4 if Cohort 3 has one DLT.
  Interventions: Drug: Lopinavir / Ritonavir
- Cohort 3: Lopinavir/Ritonavir 600mg/150mg (2 cycles) (Experimental): Cohort 3 will receive two 5-day cycles of the highest dose of the suppository (Lopinavir/Ritonavir (600mg/150mg)) in Weeks 0 and 2, if the Cohort 2 dose is safe.
  Interventions: Drug: Lopinavir / Ritonavir
- Cohort 4: Lopinavir/Ritonavir 600mg/150mg (3 cycles) (Experimental): Cohort 4 will receive three 5-day cycles of the highest dose of the suppository (Lopinavir/Ritonavir (600mg/150mg)) in Weeks 0, 2, and 4, if the Cohort 3 dose is safe.
  Interventions: Drug: Lopinavir / Ritonavir

INTERVENTIONS:
Drug: Lopinavir / Ritonavir — Human Immunodeficiency Virus (HIV) antiviral, given via suppository

SUMMARY:
This study is being done to assess the safety of lopinavir/ritonavir in patients with PLWH with AIN. 30 participants will be recruited and can expect to be on active study for approximately 3 months and long term follow up for 40 weeks.

DETAILED DESCRIPTION:
This is a Phase I modified 3 + 3 design, in which the maximum tolerated dose (MTD) will be identified. The 3 + 3 dose escalation will consist of 6 dose levels (18 participants; planned escalation described in arms below) in combination with variation in dosing schedules of the drug lopinavir/ritonavir. This design also allows for some possible intermediate doses to be examined if dose-limiting toxicities (DLTs) occur and de-escalation is needed.

An expansion cohort of 12 participants will occur at the MTD. Once the MTD is determined, then secondary outcomes will be evaluated.

Primary Objective

* To evaluate the safety and tolerability of intra-anal administration of lopinavir/ritonavir, administered via suppository with 3 different schedules, in PLWH with high-grade anal intraepithelial neoplasia (HGAIN) (AIN 2/3).

Secondary Objectives

* To measure the effect of intra-anal topical lopinavir/ritonavir administration
* To evaluate clearance of human papillomavirus (HPV)
* To elucidate the mechanism of action of protease inhibitors

ELIGIBILITY:
Inclusion Criteria:

* willing to provide informed consent
* greater than or equal to 18 years of age
* Diagnosis of biopsy-confirmed HGAIN
* Human immunodeficiency virus (HIV)-positive with CD4 count greater than 200 cells/mm^3 at screening and virologically suppressed on HIV-1 antiretroviral therapy (ART) within last 12 months
* willing to comply with all study procedures

Exclusion Criteria:

* Diagnosis of low-grade anal dysplasia (AIN, low-grade squamous intraepithelial lesion (LSIL)) by HRA.
* CD4 count less than 200 cells/mm^3 at the time of consideration for entry into the study
* unable to provide informed consent
* Pregnant or breastfeeding female
* Currently receiving systemic chemotherapy or radiation therapy for another cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) as determined by the number of participants at each dose level in the escalation cohorts who experienced a dose-limiting toxicity (DLT) | up to 5 weeks
  The MTD is the highest explored dose of lopinavir/ritonavir is the dose at which less than 33% of patients experienced a DLT. A DLT is defined as any toxicity at least possibly related to ritonavir/lopinavir with a drug-related Grade greater than or equal to 3.
Rate of Grade 3 or above Toxicities in any Organ System in the Escalation Cohorts | up to 5 weeks
  Grade 3 or above as delineated in Common Terminology Criteria for Adverse Events v 5.0 (CTCAE)

SECONDARY OUTCOMES:
Number of Participants in the Expansion Cohort Who Experience Regression of AIN2/3 Determined by Pathology | week 12, week 40
  Efficacy of intra-anal topical lopinavir/ritonavir administration determined by pathology, based on the regression of AIN2/3 at study weeks 16, 28, and 40. Regression defined as either AIN1 or no AIN lesion detected by High resolution anoscopy (HRA)/biopsy and anal cytology. Down grade of disease from AIN2/3 to AIN1 or normal.
Number of Participants in the Expansion Cohort Determined clear of HPV by PCR test | week 12, week 40
  HPV clearance determined by quantitative polymerase chain reaction (PCR) test.
Number of Tissue Samples with evidence of apoptosis measured by presence of Activated Caspase 3 | week 12, week 40
  Mechanism of action of protease inhibitors investigated with biomarker studies (immunohistochemistry and Immunofluorescence of tissue). Samples with activated caspase 3 indicate evidence of apoptosis.
Number of Tissue Samples with evidence of autophagy measured by presence of LC3β and p62 | week 12, week 40
  Mechanism of action of protease inhibitors investigated with biomarker studies (immunohistochemistry and Immunofluorescence of tissue). Samples with LC3β and p62 indicate evidence of autophagy.
Number of Tissue Samples with evidence of cellular proliferation measured by presence of Ki-67 | week 12, week 40
  Mechanism of action of protease inhibitors investigated with biomarker studies (immunohistochemistry and Immunofluorescence of tissue). Samples with Ki-67 indicate evidence of cellular proliferation.
Number of Tissue Samples with evidence of HPV positivity measured by presence of p16 | week 12, week 40
  Mechanism of action of protease inhibitors investigated with biomarker studies (immunohistochemistry and Immunofluorescence of tissue). Samples with p16 indicate evidence of HPV positivity.
Number of Tissue Samples with p53 expression | week 12, week 40
  Mechanism of action of protease inhibitors investigated with biomarker studies (immunohistochemistry and Immunofluorescence of tissue).

CONTACTS AND LOCATIONS:
Overall Officials: Evie Carchman, MD, FACS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- UW Digestive Health Center Anoscopy Clinic, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No